CLINICAL TRIAL: NCT00952705
Title: A Randomized, Partially Blind Active Controlled Study to Evaluate the Immunogenicity of MEDI8662 in Adults 18 to 49 Years of Age
Brief Title: A Study to Evaluate the Immunogenicity of Quadrivalent LAIV (MEDI8662) in Adults 18 to 49 Years of Age
Acronym: MI-CP206
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: J. A. Sliman, MD, MPH, MedImmune, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP206
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2011-12

CONDITIONS: Healthy or Stable Underlying Chronic Medical Condition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Q/LAIV-BFS (MEDI8662) (Experimental): Q/LAIV-BFS (quadrivalent influenza vaccine) (MEDI8662) was supplied in the blow-fill-seal delivery system that delivers a nominal dose of 0.2 mL into a single nostril. Each dose contained 10^7.0 ± 0.5 fluorescent focus units (FFU) of each of 4 cold-adapted, temperature-sensitive, attenuated, 6:2 reassortant influenza virus strains: A/H1N1 (A/South Dakota/6/2007), A/H3N2 (A/Uruguay/716/2007), B/Victoria (B/Malaysia/2506/2004), and B/Yamagata (B/Florida/4/2006).
  Interventions: Biological: Q/LAIV-BFS (MEDI8662)
- FluMist/B/Yamagata (Active Comparator): FluMist/B/Yamagata was administered intranasally using a Becton Dickinson Accuspray™ device. A total volume of 0.2 mL was administered intranasally (approximately 0.1 mL into each nostril). Each dose contained 10^7.0 ± 0.5 FFU of each of 3 cold-adapted, temperature-sensitive, attenuated, 6:2 reassortant influenza virus strains: A/H1N1 (A/South Dakota/6/2007), A/H3N2 (A/Uruguay/716/2007), and B/Yamagata (B/Florida/4/2006)
  Interventions: Biological: FluMist/B/Yamagata
- FluMist/B/Victoria (Active Comparator): FluMist/B/Victoria was administered intranasally using a BD Accuspray™ device. A total volume of 0.2 mL was administered intranasally (approximately 0.1 mL into each nostril). Each dose contained 10^7.0 ± 0.5 FFU of each of 3 cold-adapted, temperature-sensitive, attenuated, 6:2 reassortant influenza virus strains: A/H1N1 (A/South Dakota/6/2007), A/H3N2 (A/Uruguay/716/2007), and B/Victoria (B/Malaysia/2506/2004).
  Interventions: Biological: FluMist/B/Victoria

INTERVENTIONS:
Biological: Q/LAIV-BFS (MEDI8662) — A single dose of Q/LAIV-BFS delivered using the BFS delivery system (0.2 mL) on Day 0.
  Arms: Q/LAIV-BFS (MEDI8662)
Biological: FluMist/B/Yamagata — FluMist/B/Yamagata - 0.2 mL dose at Day 0
  Arms: FluMist/B/Yamagata
Biological: FluMist/B/Victoria — FluMist/B/Victoria - 0.2 mL dose at Day 0
  Arms: FluMist/B/Victoria

SUMMARY:
The purpose of this study was to show that quadrivalent live attenuated influenza vaccine (Q/LAIV-BFS; MEDI8662) was at least as immunogenic as two different forms of the commercial vaccine, FluMist, by comparing the strain-specific antibody levels in the blood.

DETAILED DESCRIPTION:
The primary objective of this study was to determine the immunologic noninferiority of MEDI8662, a quadrivalent live attenuated influenza vaccine (Q/LAIV) (delivered intranasally using the blow-fill-seal [BFS] delivery system) (Q/LAIV-BFS) to two trivalent formulations of licensed FluMist (delivered intranasally using the Becton Dickinson [BD] Accuspray™ device) by comparing the strain-specific geometric mean titers (GMTs) post dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 through 49 years, inclusive (reached their 18th year birthday but not yet reached their 50th year birthday) at the time of randomization
* Females of child-bearing potential, must have used an effective method of avoiding pregnancy for 30 days prior to the first dose of investigational product, and must have agreed to continue using such precautions for 60 days after the dose of investigational product. In addition, the participant must also have had a negative urine or blood pregnancy test at screening and, if screening and Day 0 do not occur on the same day, on the day of vaccination prior to randomization.
* Healthy by medical history and physical examination OR presence of stable underlying chronic medical condition for which hospitalization had not been required in the previous year

Exclusion Criteria:

* Acute illness or evidence of significant active infection at randomization
* Fever greater than or equal to 100.4 degrees F (38°C) at randomization
* History of asthma
* Any drug therapy from 15 days prior to randomization or expected drug therapy through 30 days post dose with the exception of contraceptives; topical corticosteroids or antifungals for uncomplicated dermatitis; chronic medications (including those taken on an as-needed basis) that were well tolerated and were not initiated and/or did not have a dosage change within 90 days of randomization
* Previous medical history or evidence of an intercurrent illness that may have compromised the safety of the participant in the study
* Current or expected receipt of immunosuppressive medications (inhaled and topical corticosteroids and topical calcineurin inhibitors were permitted) within a 30-day window around the dose
* Receipt of immunoglobulin or blood products within 90 days before randomization into the study or expected receipt during study participation
* Receipt of any investigational drug therapy within 30 days prior to randomization or planned receipt of any investigational drug therapy through 30 days after dosing of investigational product (use of licensed agents for indications not listed in the package insert were permitted)
* Receipt of any nonstudy vaccine within 30 days prior to randomization or planned receipt of nonstudy vaccine through 30 days after dosing
* Receipt of any influenza vaccine (investigational or licensed) in 2009 prior to randomization or anticipated receipt prior to the collection of the post-dose immunogenicity blood sample for this study
* Any known immunosuppressive condition or immune deficiency disease including known or suspected infection with human immunodeficiency virus (HIV)
* History of allergic disease or reactions likely to be exacerbated by any component of Q/LAIV-BFS including allergy to eggs, egg proteins, gentamicin, or gelatin, or serious, life threatening, or severe reactions to previous influenza vaccinations
* History of Guillain-Barré syndrome
* Use of antiviral agents with activity against influenza virus (including amantadine, rimantadine, oseltamivir and zanamivir) within 30 days prior to receipt of investigational product or anticipated use within 30 days after receipt of investigational product
* Known or suspected mitochondrial encephalomyopathy
* Pregnant or lactating female
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of participant safety or study results
* Participant, legal guardian, or immediate family member of participant who was an employee of the clinical study site or who was otherwise involved with the conduct of the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1800 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sliman, M.D., MPH, Study Director — MedImmune LLC
Locations (18):
- United States (18):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Benchmark Research, Sacramento, California
  - California Research Foundation, San Diego, California
  - Benchmark Research, San Francisco, California
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Miami Research Associates, Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Regional Clinical Research, Endwell, New York
  - Rochester Clinical Research Inc., Rochester, New York
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Benchmark Research Austin, Austin, Texas
  - Benchmark Research Ft. Worth, Fort Worth, Texas

REFERENCES:
- [Background] Sheldon EA, Jeanfreau R, Sliman JA, Charenkavanich S, Rousculp MD, Dubovsky F, Mallory RM. Immunogenicity of a quadrivalent Ann Arbor strain live attenuated influenza vaccine delivered using a blow-fill-seal device in adults: a randomized, active-controlled study*. Influenza Other Respir Viruses. 2013 Nov;7(6):1142-50. doi: 10.1111/irv.12027. Epub 2012 Oct 14. PMID 23061976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for the study within 30 days prior to randomization at investigator clinic sites in the USA. The first and last dates of informed consent were 14Aug2009 and 26Aug2009, respectively.
Pre-assignment Details: Of 1,888 participants who provided written informed consent and were screened for the study, 88 were screened but were not randomized into the study due to one or more of the following reasons: not meeting the eligibility criteria; study was full; withdrawal of consent; lost to follow-up; unable to obtain a blood sample for immunogenicity testing.
Groups:
- FluMist/B/Yamagata: FluMist/B/Yamagata was administered intranasally using a Becton Dickinson (BD) Accuspray™ device. A total volume of 0.2 mL was administered intranasally (approximately 0.1 mL into each nostril). Each dose contained 10^7.0 ± 0.5 FFU of each of 3 cold-adapted, temperature-sensitive, attenuated, 6:2 reassortant influenza virus strains: A/H1N1 (A/South Dakota/6/2007), A/H3N2 (A/Uruguay/716/2007), and B/Yamagata (B/Florida/4/2006).
Period: Overall Study
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata | FluMist/B/Victoria
Started | 1202 (Three not treated with Q/LAIV-BFS (1 treated with FluMist/B/Yamagata; 2 withdrew prior to dosing).) | 300 | 298
Completed | 1169 | 290 | 288
Not Completed | 33 | 10 | 10
Not completed — Lost to Follow-up | 24 | 8 | 9
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Death | 2 | 0 | 0
Not completed — Incarcerated post dose | 5 | 0 | 0
Not completed — Exclusion criteria not met pre dose | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata | FluMist/B/Victoria | Total
Number analyzed (Participants) | 1202 | 300 | 298 | 1800
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (9.5) | 34.0 (9.1) | 33.8 (8.8) | 33.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 701 | 169 | 167 | 1037
  Male | 501 | 131 | 131 | 763

OUTCOME MEASURES:

1. Primary Outcome: The Post Dose Strain-specific Serum Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMTs) in the Q/LAIV-BFS (MEDI8662) Arm as Compared to Those in the Combined Flumist Arms (All Flumist Group).
Description: Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% confidence intervals (CIs) for the ratios of strain-specific HAI GMTs for the specified comparisons. The GMT ratio = GMT in comparator (All FluMist group) divided by the GMT in the Q/LAIV-BFS arm.
Time Frame: Day 28 to 35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 1176 and 586 participants, respectively, received a full dose of investigational product, had a post-dose HAI measurement, and had no protocol violation that could have interfered with generation or interpretation of an immune response.
Measure: Geometric Mean (Full Range); unit: Geometric Mean Titer
Groups:
- All FluMist: All FluMist group for A/H1N1 and A/H3N2 strains, where data from both the FluMist/B/Yamagata arm and the FluMist/B/Victoria arm are combined.
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata | FluMist/B/Victoria | All FluMist
Number analyzed (Participants) | 1176 | 294 | 292 | 586
Geometric Mean Titer
  A/H1N1 | 8.1 [2 to 1448] | 7.1 [2 to 512] | 8.3 [2 to 1024] | 7.7 [2 to 1024]
  A/H3N2 | 8.3 [2 to 1024] | 8.0 [2 to 1024] | 7.4 [2 to 512] | 7.7 [2 to 1024]
  B/Yamagata | 60.3 [2 to 4096] | 54.1 [2 to 2048] | 49.8 [2 to 4096] | 51.9 [2 to 4096]
  B/Victoria | 27.4 [2 to 2048] | 19.9 [2 to 1024] | 26.7 [2 to 1024] | 23.0 [2 to 1024]
Statistical Analysis 1: Comparison: Q/LAIV-BFS (MEDI8662) vs All FluMist; Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CIs for the ratio of A/H1N1 GMTs for the specified comparison. Geometric mean titers for the A/H1N1 influenza antigen measurements were calculated as: GMT = antilog^y (mean [log^y x]) where x was the assay result and y was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV-BFS was declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for the post dose A/H1N1 GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the A/H1N1 post-dose GMT ratio: (FluMist B/Yamagata A/H1N1 + FluMist B/Victoria A/H1N1) divided by Q/LAIV-BFS A/H1N1; Bootstrapping method; Confidence intervals calculated based on bootstrapping method; Ratio of geometric mean titers = 0.95, 95% CI 2-sided [0.87 to 1.03]
Statistical Analysis 2: Comparison: Q/LAIV-BFS (MEDI8662) vs All FluMist; Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CIs for the ratio of A/H3N2 GMTs for the specified comparison. Geometric mean titers for the A/H3N2 influenza antigen measurements were calculated as: GMT = antilog^y (mean [log^y x]) where x was the assay result and y was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV-BFS was declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for the post dose A/H3N2 GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the A/H3N2 post-dose GMT ratio: (FluMist B/Yamagata A/H3N2 + FluMist B/Victoria A/H3N2) divided by Q/LAIV-BFS A/H3N2; Bootstrapping method; Confidence intervals calculated based on bootstrapping method; Ratio of geometric mean titers = 0.93, 95% CI 2-sided [0.85 to 1.00]
Statistical Analysis 3: Comparison: Q/LAIV-BFS (MEDI8662) vs FluMist/B/Yamagata; Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CIs for the ratio of B/Yamagata GMTs for the specified comparison. Geometric mean titers for the B/Yamagata influenza antigen measurements were calculated as: GMT = antilog^y (mean [log^y x]) where x was the assay result and y was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV-BFS was declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for the post dose B/Yamagata GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the B/Yamagata post-dose GMT ratio: FluMist B/Yamagata divided by Q/LAIV-BFS B/Yamagata; Bootstrapping method; Confidence intervals calculated based on bootstrapping method; Ratio of geometric mean titers = 0.90, 95% CI 2-sided [0.79 to 1.02]
Statistical Analysis 4: Comparison: Q/LAIV-BFS (MEDI8662) vs FluMist/B/Victoria; Noninferior immune response was assessed by evaluating the upper bound of the 2-sided 95% CIs for the ratio of B/Victoria GMTs for the specified comparison. Geometric mean titers for the B/Victoria influenza antigen measurements were calculated as: GMT = antilog^y (mean [log^y x]) where x was the assay result and y was the natural logarithm; Test type: Non-Inferiority or Equivalence — The immune response of Q/LAIV-BFS was declared noninferior to that of trivalent FluMist if the upper bound of the 95% CI for the post dose B/Victoria GMT ratio was ≤ 1.5. This corresponded to the statistical hypothesis of: Ho: Rj > 1.5 for any j and Ha: Rj ≤ 1.5 for all j, where Rj was the B/Victoria post-dose GMT ratio: FluMist B/Victoria divided by Q/LAIV-BFS B/Victoria; Bootstrapping method; Confidence intervals calculated based on bootstrapping method; Ratio of geometric mean titers = 0.97, 95% CI 2-sided [0.87 to 1.10]

2. Secondary Outcome: The Percentage of Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the A/H1N1 and A/H3N2 Strains in All Participants, Regardless of Baseline Serostatus.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. The comparators for seroresponse to the A/H1N1 and A/H3N2 strains were participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 1176 and 586 participants, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements for the 2 A strains, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 1176 | 586
Percentage of Participants
  A/H1N1 | 5.4 | 6.5
  A/H3N2 | 4.7 | 4.8

3. Secondary Outcome: The Percentage of Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the B/Yamagata Strain in All Participants, Regardless of Baseline Serostatus.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. The comparator for seroresponse to the B/Yamagata strain was participants in the FluMist/B/Yamagata arm.
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 300 FluMist/B/Yamagata-treated participants, 1175 and 294 participants, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements for B/Yamagata strain, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata
Number analyzed (Participants) | 1175 | 294
Percentage of Participants | 8.2 | 9.5

4. Secondary Outcome: The Percentage of Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the B/Victoria Strain in All Participants, Regardless of Baseline Serostatus.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. The comparator for seroresponse to the B/Victoria strain was participants in the FluMist/B/Victoria arm.
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 298 FluMist/B/Victoria-treated participants, 1176 and 292 participants, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements for B/Victoria strain, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Victoria
Number analyzed (Participants) | 1176 | 292
Percentage of Participants | 7.5 | 10.3

5. Secondary Outcome: The Percentage of Serosusceptible Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the A/H1N1 Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for seroresponse to the A/H1N1 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 783 and 412, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were serosusceptible to A/H1N1, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 783 | 412
Percentage of participants | 7.9 | 9.0

6. Secondary Outcome: The Percentage of Serosusceptible Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the A/H3N2 Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for seroresponse to the A/H3N2 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 746 and 386, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were serosusceptible to A/H3N2, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 746 | 386
Percentage of Participants | 6.3 | 7.0

7. Secondary Outcome: The Percentage of Serosusceptible Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the B/Yamagata Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for seroresponse to the B/Yamagata strain was participants in the FluMist/B/Yamagata arm.
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 300 FluMist/B/Yamagata-treated participants, 189 and 51, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were serosusceptible to B/Yamagata, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata
Number analyzed (Participants) | 189 | 51
Percentage of Participants | 36.0 | 35.3

8. Secondary Outcome: The Percentage of Serosusceptible Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the B/Victoria Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for seroresponse to the B/Victoria strain was participants in the FluMist/B/Victoria arm.
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 298 FluMist/B/Victoria-treated participants, 361 and 104, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were serosusceptible to B/Victoria, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Victoria
Number analyzed (Participants) | 361 | 104
Percentage of Participants | 20.8 | 26.0

9. Secondary Outcome: The Percentage of Seropositive Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the A/H1N1 Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for seroresponse to the A/H1N1 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 393 and 174, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were seropositive to A/H1N1, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 393 | 174
Percentage of participants | 0.5 | 0.6

10. Secondary Outcome: The Percentage of Seropositive Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the A/H3N2 Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for seroresponse to the A/H3N2 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 430 and 200, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were seropositive to A/H3N2, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 430 | 200
Percentage of participants | 1.9 | 0.5

11. Secondary Outcome: The Percentage of Seropositive Participants Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the B/Yamagata Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for seroresponse to the B/Yamagata strain was participants in the FluMist/B/Yamagata arm.
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 300 FluMist/B/Yamagata-treated participants, 986 and 243, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were seropositive to B/Yamagata, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata
Number analyzed (Participants) | 986 | 243
Percentage of Participants | 2.8 | 4.1

12. Secondary Outcome: The Percentage of Seropositive Subjects Experiencing Post Dose Strain-specific HAI Antibody Seroresponse to the B/Victoria Strain.
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for seroresponse to the B/Victoria strain was participants in the FluMist/B/Victoria arm.
Time Frame: Day 0 and Day 28-35
Population: Of 1199 Q/LAIV-treated and 298 FluMist/B/Victoria-treated participants, 815 and 188, respectively, received a full dose of investigational product, had pre- and post-dose HAI measurements, were seropositive to B/Victoria, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Victoria
Number analyzed (Participants) | 815 | 188
Percentage of Participants | 1.6 | 1.6

13. Secondary Outcome: The Percentage of Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the A/H1N1 and A/H3N2 Strains in All Participants, Regardless of Baseline Serostatus.
Description: The comparators to the A/H1N1 and A/H3N2 strains were participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 1176 and 586, respectively, received a full dose of investigational product, had post-dose HAI measurement for the 2 A strains, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 1176 | 586
Percentage of Participants
  A/H1N1 | 25.3 | 22.5
  A/H3N2 | 25.8 | 23.4

14. Secondary Outcome: The Percentage of Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the B/Yamagata Strain in All Participants, Regardless of Baseline Serostatus.
Description: The comparator for the B/Yamagata strain was participants in the FluMist/B/Yamagata arm.
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 300 FluMist/B/Yamagata-treated participants, 1176 and 294, respectively, received a full dose of investigational product, had post-dose HAI measurement for B/Yamagata strain, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of subjects
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata
Number analyzed (Participants) | 1176 | 294
Percentage of subjects | 78.7 | 75.2

15. Secondary Outcome: The Percentage of Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the B/Victoria Strain in All Participants, Regardless of Baseline Serostatus.
Description: The comparator for the B/Victoria strain was participants in the FluMist/B/Victoria arm.
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 298 FluMist/B/Victoria-treated participants, 1176 and 292, respectively, received a full dose of investigational product, had post-dose HAI measurement for B/Victoria strain, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Victoria
Number analyzed (Participants) | 1176 | 292
Percentage of Participants | 55.5 | 52.7

16. Secondary Outcome: The Percentage of Serosusceptible Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the A/H1N1 Strain.
Description: Participants with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for the A/H1N1 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 783 and 412, respectively, received a full dose of investigational product, had post-dose HAI measurement, were serosusceptible to A/H1N1, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 783 | 412
Percentage of participants | 2.7 | 1.7

17. Secondary Outcome: The Percentage of Serosusceptible Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the A/H3N2 Strain.
Description: Participants with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for the A/H3N2 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 746 and 386, respectively, received a full dose of investigational product, had post-dose HAI measurement, were serosusceptible to A/H3N2, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 746 | 386
Percentage of Participants | 1.5 | 1.8

18. Secondary Outcome: The Percentage of Serosusceptible Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the B/Yamagata Strain.
Description: Subjects with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for the B/Yamagata strain was participants in the FluMist/B/Yamagata arm.
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 300 FluMist/B/Yamagata-treated participants, 189 and 51, respectively, received a full dose of investigational product, had post-dose HAI measurement, were serosusceptible to B/Yamagata strain, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata
Number analyzed (Participants) | 189 | 51
Percentage of Participants | 21.7 | 19.6

19. Secondary Outcome: The Percentage of Serosusceptible Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the B/Victoria Strain.
Description: Participants with a baseline HAI titer ≤ 8 were considered to be serosusceptible for that strain. The comparator for the B/Victoria strain was participants in the FluMist/B/Victoria arm.
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 298 FluMist/B/Victoria-treated participants, 361 and 104, respectively, received a full dose of investigational product, had post-dose HAI measurement, were serosusceptible to B/Victoria strain, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Victoria
Number analyzed (Participants) | 361 | 104
Percentage of Participants | 9.7 | 13.5

20. Secondary Outcome: The Percentage of Seropositive Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the A/H1N1 Strain.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for the A/H1N1 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 393 and 174, respectively, received a full dose of investigational product, had post-dose HAI measurement, were seropositive to A/H1N1, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 393 | 174
Percentage of participants | 70.2 | 71.8

21. Secondary Outcome: The Percentage of Seropositive Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the A/H3N2 Strain.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for the A/H3N2 strain was participants in the All FluMist group (combined data for both FluMist arms).
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 598 treated participants in the All FluMist group, 430 and 200, respectively, received a full dose of investigational product, had post-dose HAI measurement, were seropositive to A/H3N2, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 430 | 200
Percentage of participants | 67.9 | 65.0

22. Secondary Outcome: The Percentage of Seropositive Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the B/Yamagata Strain.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for the B/Yamagata strain was participants in the FluMist/B/Yamagata arm.
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 300 FluMist/B/Yamagata-treated participants, 986 and 243, respectively, received a full dose of investigational product, had post-dose HAI measurement, were seropositive to B/Yamagata, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Yamagata
Number analyzed (Participants) | 986 | 243
Percentage of Participants | 89.7 | 86.8

23. Secondary Outcome: The Percentage of Seropositive Participants Achieving a Post Dose Strain-specific HAI Antibody Titer ≥ 32 to the B/Victoria Strain.
Description: Participants with a baseline HAI titer > 8 were considered to be seropositive for that strain. The comparator for the B/Victoria strain was participants in the FluMist/B/Victoria arm.
Time Frame: Day 28-35
Population: Of 1199 Q/LAIV-treated and 298 FluMist/B/Victoria-treated participants, 815 and 188, respectively, received a full dose of investigational product, had post-dose HAI measurement, were seropositive to B/Victoria, and had no protocol deviation that could have interfered with generation or interpretation of an immune response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | FluMist/B/Victoria
Number analyzed (Participants) | 815 | 188
Percentage of Participants | 75.8 | 74.5

24. Secondary Outcome: The Percentage of Participants Experiencing Each Solicited Symptom From Administration of Investigational Product Through 14 Days Post Dose
Time Frame: Days 0-14 post dose
Population: The Evaluable Safety Population for solicited symptoms included all participants who received any investigational product and had any solicited symptom data available during the reporting period.
Measure: Number; unit: Percentage of Participants
Groups:
- All FluMist: Data from both the FluMist/B/Yamagata arm and the FluMist/B/Victoria arm were combined.
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 1196 | 595
Percentage of Participants
  Any solicited symptom | 50.6 | 54.3
  Fever ≥ 100.4°F | 1.6 | 2.0
  Fever ≥ 101.3°F | 0.7 | 0.7
  Fever ≥ 102.2°F | 0.3 | 0.2
  Fever ≥ 103.1°F | 0.1 | 0.0
  Fever ≥ 104.0°F | 0.0 | 0.0
  Fever ≥ 104.9°F | 0.0 | 0.0
  Runny/stuffy nose | 31.3 | 37.6
  Sore throat | 17.3 | 15.0
  Cough | 9.6 | 7.9
  Headache | 23.8 | 24.4
  Generalized muscle aches | 8.4 | 11.1
  Decreased activity level (lethargy) or tiredness | 16.2 | 17.5
  Decreased appetite | 5.3 | 5.7

25. Secondary Outcome: The Percentage of Participants Reporting Any Adverse Event From Administration of Investigational Product Through 28 Days Post Dose
Time Frame: Days 0-28 post dose
Population: The Safety Population included participants who received any investigational product and for whom any follow-up safety data were reported.
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 1198 | 596
Percentage of Participants | 15.6 | 14.9

26. Secondary Outcome: The Percentage of Participants Reporting Any Serious Adverse Event From Administration of Investigational Product Through 28 Days Post Dose
Time Frame: Days 0-28 post dose
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 1198 | 596
Percentage of Participants | 0.3 | 0.0

27. Secondary Outcome: The Percentage of Participants Reporting Any Serious Adverse Event From Administration of Investigational Product Through 180 Days Post Dose
Time Frame: Days 0-180 post dose
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 1198 | 596
Percentage of Participants | 1.3 | 0.3

28. Secondary Outcome: The Percentage of Participants Reporting New Onset Chronic Diseases From Administration of Investigational Product Through 180 Days Post Dose
Time Frame: Days 0-180 post dose
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Number analyzed (Participants) | 1198 | 596
Percentage of Participants | 0.5 | 0.5

ADVERSE EVENTS:
Time Frame: Serious adverse events, Days 0-180 post dose; other adverse events, Days 0-28 post dose.
Description: Telephone contacts were made by site personnel to the participant at various times during the study to assess safety.
Arm/Group | Q/LAIV-BFS (MEDI8662) | All FluMist
Serious Adverse Events (participants affected / at risk) | 15/1198 | 2/596
Other Adverse Events (participants affected / at risk) | 100/1198 | 45/596
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q/LAIV-BFS (MEDI8662) (N=1198) | All FluMist (N=596)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Methycillin-resistant staphylococcal aureus test (Investigations) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q/LAIV-BFS (MEDI8662) (N=1198) | All FluMist (N=596)
Vomiting (Gastrointestinal disorders) | 6 (6) | 7 (7)
Nausea (Gastrointestinal disorders) | 14 (15) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 9 (9)
Headache (Nervous system disorders) | 16 (16) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.